CLINICAL TRIAL: NCT06671808
Title: HIV Infection Accompanied by Multi-Drug Resistant Tuberculosis: a Decadal Systematic Review and Meta-Analysis
Brief Title: HIV and Multi-Drug Resistant Tuberculosis: a Study on Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Zahedan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Kouhpayeh, Assistant Professor, Zahedan University of Medical Sciences
Other Study IDs: HIVTB2024
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: HIV Infection; MDR-TB
MeSH Terms: conditions — HIV Infections; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Examination of HIV Infection in Patients with Multi-Drug Resistant Tuberculosis (MDR-TB) — This meta-analysis examines the impact of HIV infection on the prevalence and outcomes of multi-drug resistant tuberculosis (MDR-TB) among affected populations. The analysis synthesizes data from multiple studies conducted across various countries, focusing on the correlation between HIV co-infection and MDR-TB rates, treatment outcomes, and demographic factors. The findings aim to enhance understanding of the complex interactions between HIV and MDR-TB, ultimately informing clinical practices and public health strategies.

SUMMARY:
This study aims to investigate the relationship between HIV infection and multi-drug resistant tuberculosis (MDR-TB) among affected individuals in Zahedan, Iran. It will involve a detailed analysis of patient demographics, clinical characteristics, and treatment outcomes to enhance understanding of this co-infection. The findings may inform better treatment strategies and healthcare policies for managing these diseases in similar populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 years and older) diagnosed with both HIV and multi-drug-resistant tuberculosis (MDR-TB).
* Studies published in peer-reviewed journals.
* Studies that provide data on the co-occurrence of HIV and MDR-TB.
* Participants from diverse geographical regions to enhance generalizability.
* Studies with clear definitions of MDR-TB according to WHO guidelines.

Exclusion Criteria:

* Studies that focus solely on drug-susceptible tuberculosis without MDR-TB.
* Studies involving pediatric populations (under 18 years of age).
* Non-original research such as reviews, editorials, and commentaries.
* Studies lacking sufficient data on the co-occurrence of HIV and MDR-TB.
* Studies that do not adhere to ethical guidelines for human subjects or lack appropriate ethical approvals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult individuals (aged 18 years and older) diagnosed with both HIV infection and multi-drug-resistant tuberculosis (MDR-TB). This meta-analysis synthesizes data from various studies conducted across multiple countries, including Brazil, the USA, Canada, India, Ethiopia, and several others. The population includes a diverse cohort of patients, reflecting various demographic characteristics such as age, sex, and geographical location.
  The studies included in this meta-analysis feature participants with confirmed diagnoses of HIV and MDR-TB, with a focus on understanding the co-infection dynamics, treatment outcomes, and associated health challenges. Data extraction from these studies provides insight into the prevalence and impact of MDR-TB among HIV-positive patients, highlighting the importance of tailored
Sampling Method: Non-Probability Sample
Enrollment: 222128 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of Multi-Drug Resistant Tuberculosis (MDR-TB) in HIV-Positive Patients | Data collected over the course of the studies from 2006 to 2018.
  This study aims to determine the prevalence of multi-drug resistant tuberculosis (MDR-TB) among patients co-infected with HIV. Data will be collected from various studies included in the meta-analysis, focusing on the incidence rates of MDR-TB in this population. The analysis will provide insights into the challenges faced in treating HIV-positive individuals with MDR-TB and highlight the need for targeted interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Zahedan University of Medical Sciences, Zahedan, Sistan and Baluchestan, Iran